CLINICAL TRIAL: NCT05551637
Title: Study the Efficiency of Oral Nutritional Supplementation on Nutrition Status, Digestive Disorders, Respiratory Infection and Anorexic in Children Between 24 - 71 Months Old.
Brief Title: Evaluating Oral Nutritional Supplements on Children's Nutritional Status and Digestive Health in Vietnam.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tu Nguyen Song (Other Government)
Responsible Party: Sponsor-Investigator, Tu Nguyen Song, Head of Division Planning, National Institute of Nutrition, Vietnam
Organization: National Institute of Nutrition, Vietnam (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: KAZUGOLD-NIN 176
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Undernutrition; Wasting; Malnourished
Keywords: Anorexic; Nutrition; Oral Nutritional Supplementation; Children; Digestive Condition; Nutrition Status; Wasting
MeSH Terms: conditions — Malnutrition; Cachexia; Anorexia

STUDY DESIGN:
Intervention Model Description: Step 1: Investigate the nutrition status of all children aged 24 - 71 months in 10 preschools in 10 selected communes. Expecting 3500 targets in 10 examined preschools
  Step 2: After the investigative selection, participants that meet the standard will be invited to the study ( the communes selected can be narrowed if the targets are hit). As soon as parents sign the consent paper, the study will move to the next step.
  Step 3: Groups will be divided to investigate activities. Creating a list for all participants that meet the criteria, with WHZ/BAZ <-0,5. Randomly selection based on age to ensure that there is no significant difference in the nutritional index or related indicators in the group to assess the effectiveness of the intervention (divided by class/age). Then, randomly divided the target by class into three large groups (300 targets per group)
Who Masked: Participant, Investigator
Masking Description: Control Group (311 participants): Children eat their usual dietary(not using Oral Nutritional Supplementation) for 3 months. After that, they will use the product for 3 months.
  Specific Intervention Group (311 participants): Children eat the usual dietary, with 2 glasses of Oral Nutritional Supplementation as the side meal. The product provides GOS, Calcium, Probiotics, HMO, DHA, and Taurine within 3 months of use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): (n=300): Children eat usual dietary (not using Oral Nutritional Supplementation) for 3 months. After that, they will use the product in 3 months
- specific intervention group (Experimental): (n=300): Children eat the usual dietary and use 2 glasses (49,2 gr powdered milk x 180 ml boil water/time x 2 times/day) of the Oral Nutritional Supplementation as the side meals. The product provides GOS, Calcium, Probiotics, HMO, DHA, and Taurine within 3 months of use.
  The product will be provided for subjects at school 5 days per week (From Monday to Friday) and at home on weekends.
  Interventions: Dietary Supplement: Kazu Gain Gold

INTERVENTIONS:
Dietary Supplement: Kazu Gain Gold — Kazu Gain Gold is an Oral Nutritional Supplementation made by AIWAIDO Food Joint Stock Company.
  Condition: Powder
  Color: White to light yellow
  Scent: The fresh scent of milk, gracious sugary smell.
  Date of use: 24 months from the manufactured date.
  User Manual: Mix 6 spoons of Kazu Gain Gold (equal to 49,2 grams) with 180 ml of warm water (The energy density reaches 1kal/ml). Consume 2 glasses per day or follow the directions from the medical staff. The product should consume less than 1 hour. Do not let the child eat the leftovers of the previous meal.
  Preserve: Store in a clean, dry place, and keep away from direct sunlight. Opened can or package must be closed and used up within 3 weeks.
  Arms: specific intervention group

SUMMARY:
Evaluating the efficiency of using Oral Nutritional Supplementation toward nutrition status (anthropometric index, the prevalence of wasting), digestive disorders, and anorexic in children aged 24 - 71 months.

DETAILED DESCRIPTION:
Evaluating the efficiency of using Oral Nutritional Supplementation toward the improvement of the anthropometric index (weight, height, weight for age Z-score, height for age Z-score, and weight for height Z-score ), nutrition status (the prevalence of wasting) in children aged 24 - 71 months after 3 months using the nutrient product.

Evaluating the efficiency of using Oral Nutritional Supplementation for digestive disorders and anorexic in children aged 24 - 71 months.

The research involves a randomized controlled clinical trial (RCT). The plan is expected to conduct from 2022 to 2023 with over 600 children aged 24-71 months. The nutrient product produces a high amount of energy that provides over 472kcal/100g; 15,6g/100g of protein; 20,8g/100 of fat; 55,6g/100g of carbonhydrate; 338mg/100g of alpha-Linolenic acid; 1800mg/100g of Linoleic acid; 19,7mg/100g of 2'FL HMO; 1088mg/100g of MCT; 2700mg/100g of FOS/Inulin; 55mg/100g of GOS; 1000mg/100g of Lysine; 687mg/100g of Calcium; 68mg/100g of Magnesium; 6,5mg/100g of Iron; 3,6/100g of Zinc; 41,9µg/100g of Manganese; 2176IU/100g of Vitamin A; 376 IU/100g of Vitamin D3; 44µg/100g of Vitamin K1; 820µg/100g of Vitamin B1; 900µg/100g of Vitamin B2; 610µg/100g of Vitamin B6; 1,92µg/100g Vitamin B12; 4140µg/100g of Acid Pantothenic; 115µg/100g of Acid Folic; 98,2 grams of the product, which equals 2 packs (230ml x 2 per day) will supply about 36,4% - 48,1% of the required energy for children aged 2-5 years old. Additional components include Alpha-Linolenic Acid, which provides 67% of the recommended dietary allowances (RDAs), Linolenic Acid 60, which provides 90% RDAs, and 25 other micronutrients and minerals that include some essential vitamins such as Calcium 112-114% RDAs, Iron 118-120.4% RDAs, Vitamin A 145-174% RDAs, Zinc 75-87% RDAs, Vitamin D3 62% RDAs, Seleni 53-63% RDAs, Vitamin K 63-73% RDAs, Folic Acid 76-115% RDAs. With other elements such as 2'FL HMO (19,7 mg), FOS/inulin (2700 mg), Choline ( 47 mg, Taurine 20 mg) , multi medium-chain triglyceride (MCT) (1088 mg), Bifidobacterium longum (109 CFU). The study will be conducted at schools and homes: 600 children erratically divided into 2 groups, 1 group will use the product for 3 months ( with the amount of use: twice per day, 49,2 grams each time). The product will be distributed to the students through the schools. Monitoring will be performed carefully by the commune and district Health Department and the Centers for Disease Control and Prevention weekly. The study aims to evaluate the efficiency of nutrient products toward nutrition status ( anthropometric index, the prevalence of wasting), digestive disorders, and anorexic in children aged 24-71 months.

ELIGIBILITY:
Inclusion Criteria:

* Children between the age of 24 - 71 months old that currently study in 10 preschools in the area of 10 selected communes.
* The family volunteered for the child to participate in the study
* Currently residing at 10 selected communes (over 1 year of residing)
* Z-score WHZ/BAZ < - 0.5

Exclusion Criteria:

* Lactose intolerance
* Children with a history of allergies, congenital diseases
* Intellectual disability or are suffering from acute and chronic infectious diseases

Ages: 24 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Division of Planning National Institute of Nutrition, Principal Investigator — National Institute of Nutrition, Vietnam
Locations (1):
- Yen Bai Province Obstetrics and Children's Hospital, Yên Bái, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about the organization in which this study is conducted. The Division of Planning is responsible to plan and implement the project. — http://viendinhduong.vn/en/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Location: Yen Bai Provincial Children's Hospital
  Recruitment time: August 1st, 2022
Pre-assignment Details: Subjects of the initial survey: 600 24-71-month-old children from 5 preschools of 5 communes meeting the criteria of WHZ/BAZ < -0.5 and other criteria.
  Organize training for staff on methods of collecting data, interview techniques, and nutritional status.
  Data collection implementation: The data collection schedule is notified to the District Hospital, the Provincial Center for Disease Control, and the health department of each school. Information collection sites are located at 5 schools.
Groups:
- Specific Intervention Group: (n=300): Children eat usual dietary and using 2 glasses (49,2 gr powdered milk x 180 ml boil water/time x 2 times/day) of the Oral Nutritional Supplementation as the side meals. The product provides GOS, Calcium, Probiotics, HMO, DHA, and Taurine within 3 months of use.
  The product will be provided for subjects at school in 5 days per week (From Monday to Friday) and at home on weekend.
  Kazu Gain Gold: Kazu Gain Gold is an Oral Nutritional Supplementation made by AIWAIDO Food Joint Stock Company.
  Condition: Powder
  Color: White to light yellow
  Scent: The fresh scent of milk, gracious sugary smell.
  Date of use: 24 months from the manufactured date.
  User Manual: Mix 6 spoons of Kazu Gain Gold (equal to 49,2 grams) with 180 ml of warm water (The energy density reaches 1kal/ml). Consume 2 glasses per day or follow the directions from the medical staff. The product should consume less than 1 hour. Do not let the child eat the leftovers of the previous meal.
  Preserve: Store in a clean, dry place, and keep away from direct sunlight. Opened can or package must be closed and used up within 3 weeks.
Period: Overall Study
Arm/Group | Control Group | Specific Intervention Group
Started | 300 | 300
Completed | 299 | 293
Not Completed | 1 | 7
Not completed — Lack of Efficacy | 0 | 6
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Specific Intervention Group: (n=300): Children eat the usual dietary and use 2 glasses (49.2 gr powdered milk x 180 ml boil water/time x 2 times/day) of the Oral Nutritional Supplementation as the side meals. The product provides GOS, Calcium, Probiotics, HMO, DHA, and Taurine within 3 months of use.
  The product will be provided for subjects at school 5 days per week (From Monday to Friday) and at home on weekends.
  Kazu Gain Gold: Kazu Gain Gold is an Oral Nutritional Supplement made by AIWAIDO Food Joint Stock Company.
  Condition: Powder
  Color: White to light yellow
  Scent: The fresh scent of milk, gracious sugary smell.
  Date of use: 24 months from the manufactured date.
  User Manual: Mix 6 spoons of Kazu Gain Gold (equal to 49.2 grams) with 180 ml of warm water (The energy density reaches 1kal/ml). Consume 2 glasses per day or follow the directions from the medical staff. The product should consume less than 1 hour. Do not let the child eat the leftovers of the previous meal.
  Preserve: Store in a clean, dry place, and avoid direct sunlight. Opened can or package must be closed and used up within 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Control Group | Specific Intervention Group | Total
Number analyzed (Participants) | 299 | 293 | 592
Age, Customized [Count of Participants; unit: Participants]
  Age group (by months old): 24 - 35.9 months | 52 | 40 | 92
  Age group (by months old): 36 - 47.9 months | 68 | 82 | 150
  Age group (by months old): 48 - 59.9 months | 97 | 104 | 201
  Age group (by months old): 60 - 71.9 months | 82 | 67 | 149
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 141 | 291
  Male | 149 | 152 | 301
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Schools: Cam Nhan | 61 | 67 | 128
  Schools: Tan Nguyen | 43 | 65 | 108
  Schools: Vinh Kien | 55 | 44 | 99
  Schools: Vu Linh | 63 | 59 | 122
  Schools: Yen Thanh | 77 | 58 | 135
Anthropometric characteristics of the subjects at the time of initial investigation [Mean (Standard Deviation); unit: Z-score]
  Z-Score Weight for age | -1.66 (0.69) | -1.67 (0.67) | -1.66 (0.68)
  Z-Score Height for age | -1.31 (0.86) | -1.36 (0.79) | -1.33 (0.82)
  Z-Score Weight for height | -1.32 (0.58) | -1.30 (0.60) | -1.31 (0.59)
Weight [Mean (Standard Deviation); unit: kilograms] | 13.43 (1.99) | 13.42 (2.05) | 13.425 (2.02)
Height [Mean (Standard Deviation); unit: centimeters] | 98.34 (7.86) | 98.13 (7.48) | 98.2 (7.67)
Months of age [Mean (Standard Deviation); unit: months] | 50.4 (12.3) | 50.3 (11.5) | 50.35 (11.9)

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Digestive Disorders and Anorexia Nervosa
Description: Children in intervention group will have more improvement in the digestive disorders and anorexic than children control group
Time Frame: From date of using the product until the date of first documented improvement, assessed up to 3 months
Measure: Number; unit: participants
Groups:
- Specific Intervention Group: (n=300): Children eat the usual dietary and use 2 glasses (49,2 gr powdered milk x 180 ml boil water/time x 2 times/day) of the Oral Nutritional Supplementation as the side meals. The product provides GOS, Calcium, Probiotics, HMO, DHA, and Taurine within 3 months of use.
  The product will be provided for subjects at school 5 days per week (From Monday to Friday) and at home on weekends.
  Kazu Gain Gold: Kazu Gain Gold is an Oral Nutritional Supplement made by AIWAIDO Food Joint Stock Company.
  Condition: Powder
  Color: White to light yellow
  Scent: The fresh scent of milk, gracious sugary smell.
  Date of use: 24 months from the manufactured date.
  User Manual: Mix 6 spoons of Kazu Gain Gold (equal to 49,2 grams) with 180 ml of warm water (The energy density reaches 1kal/ml). Consume 2 glasses per day or follow the directions from the medical staff. The product should consume less than 1 hour. Do not let the child eat the leftovers of the previous meal.
  Preserve: Store in a clean, dry place, and avoid direct sunlight. Opened can or package must be closed and used up within 3 weeks.
Arm/Group | Control Group | Specific Intervention Group
Number analyzed (Participants) | 299 | 293
participants
  Before intervention (T0) | 219 | 212
  After 3 months | 175 | 155

2. Primary Outcome: Change in Weight (kg)
Description: Weight is measured in kg with one decimal value by the Body composition analyzer TANITA scale. The scale is checked and adjusted before use. Children wear light clothing, remove shoes and sandals, and sit or lie balanced at the centre of the scale. When the balance is stable, read and write the result in kg and an odd number after the comma.
  All data will be measured at the time T0 (at baseline) and T3 (after 3 months)
Time Frame: over 1 and 3 months
Population: The classified population contains children who had consumed more than 75% of the amount of assigned milk and participated 90% during study time, with enough data on height and weight and interview forms from both assessments to be included in the analysis of the results.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Control Group | Specific Intervention Group
Number analyzed (Participants) | 299 | 298
kilograms
  Before intervention (T0) | 13.43 (1.99) | 13.5 (2.08)
  After 1 month (T1) | 13.77 (2.06) | 14.04 (2.19)
  After 2 months (T2) | 14.09 (2.03) | 14.35 (2.20)
  After 3 months (T3) | 14.24 (2.03) | 14.52 (2.23)
  Difference between T1 - T0 | 0.35 (0.46) | 0.54 (0.52)
  Difference between T2 - T0 | 0.66 (0.54) | 0.85 (0.59)
  Difference between T3 - T0 | 0.81 (0.53) | 1.01 (0.65)

3. Primary Outcome: Change of Weight for Age Z-score
Description: Change of average weight for age Z Score using the World's Health Organization (WHO) software Anthro and WHO AnthroPlus. Moreover, compare the difference between before intervention and after the intervention. A Z-score of 0 represents the population median. The standard deviations above the median represent a better outcome and vice versa.
Time Frame: over 1 and 3 months
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: Z-score
Arm/Group | Control Group | Specific Intervention Group
Number analyzed (Participants) | 299 | 298
Z-score
  Before intervention (T0) | -1.66 (0.70) | -1.62 (0.73)
  After 1 month (T1) | -1.58 (0.70) | -1.44 (0.79)
  After 2 months (T2) | -1.47 (0.70) | -1.34 (0.77)
  After 3 months (T3) | -1.47 (0.71) | -1.33 (0.79)
  Difference between T1 - T0 | 0.07 (0.27) | 0.18 (0.31)
  Difference between T2 - T0 | 0.18 (0.31) | 0.28 (0.33)
  Difference between T3 - T0 | 0.19 (0.31) | 0.29 (0.35)

4. Primary Outcome: Change of Weight for Height Z-score
Description: Change of average weight for height Z Score using WHO Anthro and WHO AnthroPlus. Moreover, compare the difference between before intervention and after the intervention. A Z-score of 0 represents the population median. The standard deviations above the median represent a better outcome and vice versa.
Time Frame: over 1 and 3 months
Population: Change of average weight for height Z Score and the difference between before intervention and after the intervention
Measure: Median (Standard Deviation); unit: Z-score
Arm/Group | Control Group | Specific Intervention Group
Number analyzed (Participants) | 299 | 298
Z-score
  Before intervention (T0) | -1.32 (0.58) | -1.32 (0.60)
  After 1 month (T1) | -1.13 (0.61) | -0.98 (0.68)
  After 2 months (T2) | -1.03 (0.62) | -0.89 (0.66)
  After 3 months (T3) | -0.96 (0.60) | -0.84 (0.66)
  Difference between T1 - T0 | 0.19 (0.40) | 0.35 (0.47)
  Difference between T2 - T0 | 0.29 (0.45) | 0.43 (0.51)
  Difference between T3 - T0 | 0.36 (0.46) | 0.48 (0.53)

5. Primary Outcome: Change in Height (cm)
Description: A wooden stadiometer measures height by precisely 0.1cm. Children stand up straight, their eyes look straight, and the top of their head touches the wooden shelf fixed at a 0 cm position. The child's whole body ensures that 9 points touch the surface of the ruler: occipital, shoulder blade, buttocks, calf, and heel. The result is recorded in cm and an odd number after the comma.
  All data will be measured at the time T0 (at baseline) and T3 (after 3 months)
Time Frame: over 1 and 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Control Group | Specific Intervention Group
Number analyzed (Participants) | 299 | 298
centimeters
  Before intervention (T0) | 98.34 (7.86) | 98.62 (7.86)
  After 1 month (T1) | 98.88 (7.89) | 99.14 (7.88)
  After 2 months (T2) | 99.68 (7.72) | 99.96 (7.92)
  After 3 months (T3) | 99.95 (7.77) | 100.35 (7.88)
  Difference between T1 - T0 | 0.54 (0.72) | 0.52 (0.69)
  Difference between T2 - T0 | 1.32 (0.82) | 1.34 (0.75)
  Difference between T3 - T0 | 1.61 (0.84) | 1.73 (0.85)

6. Primary Outcome: Change of Height for Age Z-score
Description: Change of average height for age Z Score using WHO Anthro and WHO AnthroPlus. Moreover, compare the difference between before intervention and after the intervention. A Z-score of 0 represents the population median. The standard deviations above the median represent a better outcome and vice versa.
Time Frame: over 1 and 3 months
Population: Change of average weight for age Z Score and the difference between before intervention and after the intervention
Measure: Median (Standard Deviation); unit: Z-score
Arm/Group | Control Group | Specific Intervention Group
Number analyzed (Participants) | 299 | 298
Z-score
  Before intervention (T0) | -1.31 (0.86) | -1.24 (0.94)
  After 1 month (T1) | -1.38 (0.85) | -1.32 (0.93)
  After 2 months (T2) | -1.30 (0.84) | -1.24 (0.93)
  After 3 months (T3) | -1.36 (0.85) | -1.27 (0.94)
  Difference between T1 - T0 | -0.07 (0.18) | -0.07 (0.17)
  Difference between T2 - T0 | 0.01 (0.19) | 0.00 (0.19)
  Difference between T3 - T0 | -0.05 (0.20) | -0.03 (0.21)

7. Secondary Outcome: Changes in the Rate of Children Have Gastrointestinal Diseases
Description: Changes in the percentage of anorexia, the incidence of gastrointestinal diseases (diarrhea, constipation) after intervention
Time Frame: over 1 and 3 months
Measure: Number; unit: participants
Arm/Group | Control Group | Specific Intervention Group
Number analyzed (Participants) | 299 | 293
participants
  Have diarrhea: During the first month of intervention (T1) | 3 | 11
  Have diarrhea: During the second month of intervention (T2) | 5 | 3
  Have diarrhea: During the third month of intervention (T3) | 4 | 1
  Have constipation: During the first month of intervention (T1) | 0 | 0
  Have constipation: During the second month of intervention (T2) | 0 | 0
  Have constipation: During the third month of intervention (T3) | 1 | 0

8. Secondary Outcome: Changes in the Rate of Malnutrition and Risk of Underweight, Stunting and Wasting
Description: Changes in the rate of malnutrition and risk of underweight, wasting and stunting after 1, 2 and 3 months of intervention
Time Frame: over 1 and 3 months
Measure: Number; unit: participants
Arm/Group | Control Group | Specific Intervention Group
Number analyzed (Participants) | 299 | 293
participants
  Malnutrition and risk of underweight : Before intervention (T0) | 246 | 244
  Malnutrition and risk of underweight : After 1 month (T1) | 240 | 226
  Malnutrition and risk of underweight : After 2 months (T2) | 221 | 207
  Malnutrition and risk of underweight : After 3 months (T3) | 220 | 209
  Malnutrition and risk of stunting : Before intervention (T0) | 187 | 205
  Malnutrition and risk of stunting : After 1 month (T1) | 196 | 208
  Malnutrition and risk of stunting : After 2 months (T2) | 184 | 206
  Malnutrition and risk of stunting : After 3 months (T3) | 191 | 204
  Malnutrition and risk of wasting : Before intervention (T0) | 197 | 187
  Malnutrition and risk of wasting : After 1 month (T1) | 169 | 146
  Malnutrition and risk of wasting : After 2 months (T2) | 148 | 127
  Malnutrition and risk of wasting : After 3 months (T3) | 129 | 118

ADVERSE EVENTS:
Time Frame: At school, the intervention product would passed to teachers (on weekdays) and parents (at weekends). The oral product should be used every day based on the instructions. Observe the participants every day and note down any situation that occurred in the designed notebook. This will continue every day for three months.
Description: Adverse events were recorded along with health status, product usage, abnormal symptoms, and daily health conditions in a monitoring log maintained by parents and teachers under the supervision of healthcare staff and community health officers at the district level.
  Collaborators are responsible for advising research subjects or requesting to go to a medical facility when experiencing nausea, diarrhea or other unusual symptoms
Arm/Group | Control Group | Specific Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/299 | 0/293
Serious Adverse Events (participants affected / at risk) | 0/299 | 0/293
Other Adverse Events (participants affected / at risk) | 0/299 | 0/293

LIMITATIONS AND CAVEATS:
Due to research ethics, the intervention and control groups consume the products. Moreover, some children might drink other supplements or products that improve their weight and height at home. However, it does not strongly affect the result of this research

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT05551637/Prot_SAP_000.pdf